CLINICAL TRIAL: NCT00005860
Title: A Phase I Study of Intraperitoneal Oxaliplatin Alone and in Combination With Intraperitoneal Floxuridine and Leucovorin in Patients With Advanced Metastatic Cancer Confined to the Peritoneal Cavity
Brief Title: Oxaliplatin With Or Without Floxuridine and Leucovorin in Treating Patients With Metastatic Cancer of the Peritoneum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067890; MSKCC-99100; NCI-T99-0107
Record Dates: First submitted 2000-06-02; First posted 2004-04-02 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2002-05

CONDITIONS: Cancer
Keywords: stage IV colon cancer; stage IV gastric cancer; recurrent gastric cancer; recurrent pancreatic cancer; recurrent colon cancer; regional neuroblastoma; stage 4S neuroblastoma; recurrent neuroblastoma; regional gastrointestinal carcinoid tumor; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; advanced adult primary liver cancer; recurrent adult primary liver cancer; gastrinoma; small intestine adenocarcinoma; small intestine lymphoma; small intestine leiomyosarcoma; unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; insulinoma; recurrent islet cell carcinoma; WDHA syndrome; somatostatinoma; pancreatic polypeptide tumor; glucagonoma; regional pheochromocytoma; metastatic pheochromocytoma; recurrent pheochromocytoma; extragonadal germ cell tumor; liver metastases; malignant ascites; newly diagnosed carcinoma of unknown primary; carcinoma of the appendix; pseudomyxoma peritonei; fallopian tube cancer; primary peritoneal cavity cancer; recurrent carcinoma of unknown primary; gastrointestinal stromal tumor; stage IV pancreatic cancer
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Neuroblastoma; Carcinoma, Hepatocellular; Gastrinoma; Gallbladder Neoplasms; Bile Duct Neoplasms; Insulinoma; Carcinoma, Islet Cell; Vipoma; Somatostatinoma; Glucagonoma; Pheochromocytoma; Appendiceal Neoplasms; Pseudomyxoma Peritonei; Fallopian Tube Neoplasms; Neoplasms, Unknown Primary; Gastrointestinal Stromal Tumors | interventions — Floxuridine; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: floxuridine
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of oxaliplatin with or without floxuridine and leucovorin in treating patients who have metastatic cancer of the peritoneum.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of intraperitoneal oxaliplatin with or without intraperitoneal floxuridine and leucovorin calcium in patients with metastatic cancer confined to the peritoneal cavity.
* Determine dose limiting and nondose limiting toxicities and pharmacokinetics of these treatment regimens in this patient population.

OUTLINE: This is a dose escalation study of oxaliplatin.

Patients receive intraperitoneal (IP) oxaliplatin over 1 hour on day 1 every 2 weeks for 2 courses.

Beginning at course 3, patients receive oxaliplatin with floxuridine and leucovorin calcium IP on day 1 and floxuridine and leucovorin calcium IP alone on days 2 and 3. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients with complete surgical resection of disease receive a total of 6 courses of combination chemotherapy.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: A total of 3-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic or unresectable cancer largely confined to the peritoneal cavity

  * Fully resected and/or electrocauterized metastatic disease involving the peritoneum (stage IV, no residual disease) allowed
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* SGOT/SGPT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* No history of allergy to platinum compounds or antiemetics that would preclude study
* No other uncontrolled illness (e.g., active infection)
* No evidence of neuropathy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior cytotoxic chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics

Other:

* No other concurrent investigational agents
* No concurrent antiretroviral therapy (HAART)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B. Saltz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States